CLINICAL TRIAL: NCT02434159
Title: Role of Cardiac Computed Tomography and Cardiac Magnetic Resonance in Optimising Response to Cardiac Resynchronisation Therapy
Brief Title: Role of Cardiac Computed Tomography in Optimising Response to Cardiac Resynchronisation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/0583
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

ARMS (2):
- Scan (Active Comparator): Heart scan prior to device insertion
  Interventions: Other: Heart scan
- No scan (No Intervention): No heart scan prior to device insertion

INTERVENTIONS:
Other: Heart scan
  Arms: Scan

SUMMARY:
The purpose of this study is to determine if detailed scanning of the heart before biventricular device insertion will improve outcomes for heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18, <90
2. Patients with moderate or severe heart failure ( NYHA functional class II-IV) due to ischaemic or non-ischaemic cardiomyopathy.
3. QRS duration >120ms on 12 lead ECG
4. LVEF < 35%
5. LVEDD >55 mm
6. Patients on optimum medical treatment for heart failure. The doses of these medications have been stable for 3 months.

Exclusion Criteria:

1. Patients with a cardiac or cerebral ischemic event within the previous three months prior to recruitment
2. Patients who had had an atrial arrhythmia within one month prior to recruitment
3. Patients with a systolic blood pressure of more than 170 or less than 80 mm Hg
4. Patients with a heart rate of more than 140 beats per minute
5. Patients with severe renal failure (eGFR < 30)
6. Patients with a history of allergy to iodine based contrast agents
7. Predicted life expectancy < 1 year
8. Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom